CLINICAL TRIAL: NCT02735395
Title: Impact of Different Dosages and Time of Administration of Metronidazole and Amoxicillin in the Treatment of Generalized Chronic Periodontitis: A Randomized Clinical Trial
Brief Title: Dose and Duration of Metronidazole and Amoxicillin for Treatment of Chronic Periodontitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Belén Retamal-Valdes, DDS, MSc, PhD Student, University of Guarulhos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SISNEP/513
Record Dates: First submitted 2016-03-22; First posted 2016-04-12 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Chronic Periodontitis
Keywords: Periodontal Diseases; Metronidazole; Amoxicillin; Chronic periodontitis; Root Planing
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (Placebo Comparator): Scaling and root planing (SRP) + two placebo pills thrice a day (TID) for 14 days (control group)
  Interventions: Procedure: Scaling and root planing (SRP); Other: Placebo 400 (14 days); Other: Placebo 500
- MTZ 250 (7 days) (Active Comparator): SRP + MTZ (250mg/TID) + AMX, for 7 days and placebos for another 7 days
  Interventions: Procedure: Scaling and root planing (SRP); Drug: Metronidazole 250 (7 days); Drug: Amoxicillin; Other: Placebo 250 (7 days)
- MTZ 400 (7 days) (Active Comparator): SRP + MTZ (400mg/TID) + AMX, for 7 days and placebos for another 7 days
  Interventions: Procedure: Scaling and root planing (SRP); Drug: Metronidazole 400 (7 days); Drug: Amoxicillin; Other: Placebo 400 (7 days)
- MTZ 250 (14 days) (Active Comparator): SRP +MTZ (250mg/TID) + AMX for 14 days
  Interventions: Procedure: Scaling and root planing (SRP); Drug: Metronidazole 250 (14 days); Drug: Amoxicillin
- MTZ 400 (14 days) (Active Comparator): SRP +MTZ (400mg/TID) + AMX for 14 days
  Interventions: Procedure: Scaling and root planing (SRP); Drug: Metronidazole 400 (14 days); Drug: Amoxicillin

INTERVENTIONS:
Procedure: Scaling and root planing (SRP) — SRP performed in four to six appointments lasting approximately 1 h each, using manual curettes (Hu-Friedy, Chicago, IL, USA) and ultrasonic device (Cavitron Select SPC, Dentsply professional, York, PA, USA) under local anesthesia. The deep sites will be scaled throughout the first week and treatment of the entire oral cavity will be completed in 14 days.
Drug: Metronidazole 250 (7 days) — Subjects will intake Metronidazole 250 mg. for 7 days, starting immediately after the first session of Scaling and Root Planing.
  Arms: MTZ 250 (7 days)
Drug: Metronidazole 400 (7 days) — Subjects will intake Metronidazole 400 mg. for 7 days, starting immediately after the first session of Scaling and Root Planing.
  Arms: MTZ 400 (7 days)
Drug: Metronidazole 250 (14 days) — Subjects will intake Metronidazole 250 mg. for 14 days, starting immediately after the first session of Scaling and Root Planing.
  Arms: MTZ 250 (14 days)
Drug: Metronidazole 400 (14 days) — Subjects will intake Metronidazole 400 mg. for 14 days, starting immediately after the first session of Scaling and Root Planing.
  Arms: MTZ 400 (14 days)
Drug: Amoxicillin — Subjects will intake Amoxicillin 500 mg. for 14 days, starting immediately after and the first session of Scaling and Root Planing.
  Arms: MTZ 250 (14 days); MTZ 250 (7 days); MTZ 400 (14 days); MTZ 400 (7 days)
Other: Placebo 250 (7 days) — Subjects will intake placebo of Metronidazole 250 mg. for 7 days, starting immediately after to intake Metronidazole 250 mg.
  Arms: MTZ 250 (7 days)
Other: Placebo 400 (7 days) — Subjects will intake placebo of Metronidazole 400 mg. for 7 days, starting immediately after to intake Metronidazole 400 mg.
  Arms: MTZ 400 (7 days)
Other: Placebo 400 (14 days) — Subjects will intake placebo of Metronidazole 400 mg. for 14 days, starting immediately after the first session of Scaling and Root Planing.
  Arms: Control
Other: Placebo 500 — Subjects will intake placebo of Amoxicillin 500 mg. for 14 days, starting immediately after the first session of Scaling and Root Planing.
  Arms: Control

SUMMARY:
The aim of this study was to compare the clinical and microbiological outcomes of different dosages of metronidazole (MTZ) and of the duration of the systemic administration of MTZ and amoxicillin as adjunct to scaling and root planing (SRP) in the treatment of generalized chronic periodontitis (GChP).

DETAILED DESCRIPTION:
Randomized clinical trials and systematic reviews have shown that the use of the combination of metronidazole (MTZ) and amoxicillin (AMX) significantly improves the benefits of the SRP in the treatment of subjects with periodontitis. However, the optimal dosage and interval of administration of these antibiotics are still unclear. Therefore, the aim of this study was to compare the clinical and microbiological outcomes of different dosages and duration of the systemic administration of the combination of MTZ and AMX as adjunct to scaling and root planing (SRP) in the treatment of generalized chronic periodontitis (GChP). One hundred ten subjects will be randomly assigned to receive SRP plus placebo, or SRP combined with 250 mg or 400 mg of MTZ, plus AMX (500 mg) TID, for either 7 or 14 days. Subjects will be clinically and microbiologically monitored up to 1 year post-therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥30 years of age;
* at least 15 teeth (excluding third molars and teeth with advanced decay indicated for extraction)
* a minimum of 6 teeth with at least one site each with probing depth (PD) and clinical * attachment level (CAL) ≥5 mm;
* at least 30% of the sites with PD and CAL ≥4 mm and bleeding on probing (BOP).

Exclusion Criteria:

* pregnancy
* breastfeeding
* current smoking and former smoking within the past 5 years;
* systemic diseases that could affect the progression of periodontitis (e.g. diabetes, immunological disorders, osteoporosis);
* scaling and root planing an in the previous 12 months;
* antibiotic therapy in the previous 6 months;
* long-term intake of anti-inflammatory medications;
* need for antibiotic pre-medication for routine dental therapy;
* allergy to metronidazole and/or amoxicillin.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-07; Primary Completion 2014-05 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects reaching ≤ 4 periodontal sites with probing depth (PD) ≥ 5 mm at 12 months | 12 months

SECONDARY OUTCOMES:
Number of sites with PD ≥ 5 mm | Baseline, 3, 6 and 12 months
Number of sites with PD ≥ 6 mm | Baseline, 3, 6 and 12 months
Number of sites with PD ≥ 7 mm | Baseline, 3, 6 and 12 months
Reduction in the number of sites with PD ≥ 5 mm | Baseline, 3, 6 and 12 months
Reduction in the number of sites with PD ≥ 6 mm | Baseline, 3, 6 and 12 months
Reduction in the number of sites with PD ≥ 7 mm | Baseline, 3, 6 and 12 months
Full-mouth PD | Baseline, 3, 6 and 12 months
Full-mouth clinical attachment level | Baseline, 3, 6 and 12 months
Percentage of sites with bleeding on probing | Baseline, 3, 6 and 12 months
Percentage of sites with plaque accumulation | Baseline, 3, 6 and 12 months
Percentage of sites with marginal bleeding | Baseline, 3, 6 and 12 months
Occurrence of headache obtained through a questionnaire of adverse effects | 14 days after the beginning of treatments
Occurrence of vomiting obtained through a questionnaire of adverse effects | 14 days after the beginning of treatments
Occurrence of diarrhea obtained through a questionnaire of adverse effects | 14 days after the beginning of treatments
Occurrence of metallic taste obtained through a questionnaire of adverse effects | 14 days after the beginning of treatments
Occurrence of nausea obtained through a questionnaire of adverse effects | 14 days after the beginning of treatments
Occurrence of irritability obtained through a questionnaire of adverse effects | 14 days after the beginning of treatments
Proportions of periodontal pathogenic bacterial species | Baseline, 3, 6 and 12 months
Counts of periodontal pathogenic bacterial species | Baseline, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Magda Feres, Professor, Study Chair — Guarulhos University
Locations (1):
- Guarulhos University, Guarulhos, São Paulo, Brazil

REFERENCES:
- [Background] Aimetti M, Romano F, Guzzi N, Carnevale G. Full-mouth disinfection and systemic antimicrobial therapy in generalized aggressive periodontitis: a randomized, placebo-controlled trial. J Clin Periodontol. 2012 Mar;39(3):284-94. doi: 10.1111/j.1600-051X.2011.01795.x. Epub 2012 Jan 4. PMID 22220822
- [Background] Carvalho LH, D'Avila GB, Leao A, Haffajee AD, Socransky SS, Feres M. Scaling and root planing, systemic metronidazole and professional plaque removal in the treatment of chronic periodontitis in a Brazilian population. I. clinical results. J Clin Periodontol. 2004 Dec;31(12):1070-6. doi: 10.1111/j.1600-051X.2004.00605.x. PMID 15560807
- [Background] Cionca N, Giannopoulou C, Ugolotti G, Mombelli A. Amoxicillin and metronidazole as an adjunct to full-mouth scaling and root planing of chronic periodontitis. J Periodontol. 2009 Mar;80(3):364-71. doi: 10.1902/jop.2009.080540. PMID 19254119
- [Background] Feres M, Figueiredo LC, Soares GM, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015 Feb;67(1):131-86. doi: 10.1111/prd.12075. PMID 25494600
- [Background] Feres M, Soares GM, Mendes JA, Silva MP, Faveri M, Teles R, Socransky SS, Figueiredo LC. Metronidazole alone or with amoxicillin as adjuncts to non-surgical treatment of chronic periodontitis: a 1-year double-blinded, placebo-controlled, randomized clinical trial. J Clin Periodontol. 2012 Dec;39(12):1149-58. doi: 10.1111/jcpe.12004. Epub 2012 Sep 27. PMID 23016867
- [Background] Guerrero A, Griffiths GS, Nibali L, Suvan J, Moles DR, Laurell L, Tonetti MS. Adjunctive benefits of systemic amoxicillin and metronidazole in non-surgical treatment of generalized aggressive periodontitis: a randomized placebo-controlled clinical trial. J Clin Periodontol. 2005 Oct;32(10):1096-107. doi: 10.1111/j.1600-051X.2005.00814.x. PMID 16174275
- [Background] Mestnik MJ, Feres M, Figueiredo LC, Soares G, Teles RP, Fermiano D, Duarte PM, Faveri M. The effects of adjunctive metronidazole plus amoxicillin in the treatment of generalized aggressive periodontitis: a 1-year double-blinded, placebo-controlled, randomized clinical trial. J Clin Periodontol. 2012 Oct;39(10):955-61. doi: 10.1111/j.1600-051X.2012.01932.x. Epub 2012 Aug 6. PMID 22882646
- [Background] Mestnik MJ, Feres M, Figueiredo LC, Duarte PM, Lira EA, Faveri M. Short-term benefits of the adjunctive use of metronidazole plus amoxicillin in the microbial profile and in the clinical parameters of subjects with generalized aggressive periodontitis. J Clin Periodontol. 2010 Apr;37(4):353-65. doi: 10.1111/j.1600-051X.2010.01538.x. PMID 20447259
- [Background] Miranda TS, Feres M, Perez-Chaparro PJ, Faveri M, Figueiredo LC, Tamashiro NS, Bastos MF, Duarte PM. Metronidazole and amoxicillin as adjuncts to scaling and root planing for the treatment of type 2 diabetic subjects with periodontitis: 1-year outcomes of a randomized placebo-controlled clinical trial. J Clin Periodontol. 2014 Sep;41(9):890-9. doi: 10.1111/jcpe.12282. Epub 2014 Jul 17. PMID 24930639
- [Background] Rabelo CC, Feres M, Goncalves C, Figueiredo LC, Faveri M, Tu YK, Chambrone L. Systemic antibiotics in the treatment of aggressive periodontitis. A systematic review and a Bayesian Network meta-analysis. J Clin Periodontol. 2015 Jul;42(7):647-57. doi: 10.1111/jcpe.12427. PMID 26087839
- [Background] Sgolastra F, Gatto R, Petrucci A, Monaco A. Effectiveness of systemic amoxicillin/metronidazole as adjunctive therapy to scaling and root planing in the treatment of chronic periodontitis: a systematic review and meta-analysis. J Periodontol. 2012 Oct;83(10):1257-69. doi: 10.1902/jop.2012.110625. Epub 2012 Feb 14. PMID 22220767
- [Background] Sgolastra F, Petrucci A, Gatto R, Monaco A. Effectiveness of systemic amoxicillin/metronidazole as an adjunctive therapy to full-mouth scaling and root planing in the treatment of aggressive periodontitis: a systematic review and meta-analysis. J Periodontol. 2012 Jun;83(6):731-43. doi: 10.1902/jop.2011.110432. Epub 2011 Nov 3. PMID 22050545
- [Background] Silva MP, Feres M, Sirotto TA, Soares GM, Mendes JA, Faveri M, Figueiredo LC. Clinical and microbiological benefits of metronidazole alone or with amoxicillin as adjuncts in the treatment of chronic periodontitis: a randomized placebo-controlled clinical trial. J Clin Periodontol. 2011 Sep;38(9):828-37. doi: 10.1111/j.1600-051X.2011.01763.x. Epub 2011 Jul 15. PMID 21762197
- [Background] Zandbergen D, Slot DE, Niederman R, Van der Weijden FA. The concomitant administration of systemic amoxicillin and metronidazole compared to scaling and root planing alone in treating periodontitis: =a systematic review=. BMC Oral Health. 2016 Feb 29;16:27. doi: 10.1186/s12903-015-0123-6. PMID 26928597
- [Background] Zandbergen D, Slot DE, Cobb CM, Van der Weijden FA. The clinical effect of scaling and root planing and the concomitant administration of systemic amoxicillin and metronidazole: a systematic review. J Periodontol. 2013 Mar;84(3):332-51. doi: 10.1902/jop.2012.120040. Epub 2012 May 21. PMID 22612369
- [Background] Soares GM, Mendes JA, Silva MP, Faveri M, Teles R, Socransky SS, Wang X, Figueiredo LC, Feres M. Metronidazole alone or with amoxicillin as adjuncts to non-surgical treatment of chronic periodontitis: a secondary analysis of microbiological results from a randomized clinical trial. J Clin Periodontol. 2014 Apr;41(4):366-76. doi: 10.1111/jcpe.12217. PMID 24834504
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- [Derived] Borges I, Faveri M, Figueiredo LC, Duarte PM, Retamal-Valdes B, Montenegro SCL, Feres M. Different antibiotic protocols in the treatment of severe chronic periodontitis: A 1-year randomized trial. J Clin Periodontol. 2017 Aug;44(8):822-832. doi: 10.1111/jcpe.12721. Epub 2017 Jul 26. PMID 28303587